CLINICAL TRIAL: NCT06090357
Title: Biomechanical Functional Evaluation of Plantar Pressures After Foot and Ankle Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PresP
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Plantar Pressure
Keywords: foot; ankle; Post-operative; plantar pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-surgical foot and ankle patients (Experimental)
  Interventions: Other: Plantar pressure

INTERVENTIONS:
Other: Plantar pressure — Biomechanical functional assessments investigate specific variables: gait analysis, stabilometry, kinematics and kinetics of joint movements, activation, and strength of specific muscle groups.

SUMMARY:
The described surgical techniques for the treatment of foot and ankle pathologies are numerous. In order to objectively assess the outcomes of these procedures, evaluation methods are typically used, primarily considering pain symptoms, residual functionality, the correction of any deformities achieved, and radiographic parameters. Conversely, assessments of plantar pressures, as a potential indicator of functional and biomechanical recovery, are still not widely utilized. Biomechanical functional assessments examine specific variables, including gait analysis, stabilometry, kinematics and kinetics of joint movements, and the activation and strength of particular muscle groups. These assessments can be conducted by specialized personnel using dedicated equipment such as a baropodometric platform and inertial sensors.

This study aims to, for the first time in the literature, present the results related to plantar pressures from different surgical treatments of the foot and ankle

ELIGIBILITY:
Inclusion Criteria:

* Patients who need to undergo surgical intervention
* Patients of both sexes aged between 18-75 years
* Patients who have provided their written informed consent to participate in the study
* Patients who have expressed their willingness to attend the Institute for the 6-month follow-up

Exclusion Criteria:

* Patients with severe postural instability
* Patients with cognitive deficits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | At baseline (day 0)
  Visual Analogue Scale (VAS) is one of the pain rating scales. It is unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).
Visual Analogue Scale | After 6 months
  Visual Analogue Scale (VAS) is one of the pain rating scales. It is unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giannini S. Kenneth A. Johnson Memorial Lecture. Operative treatment of the flatfoot: why and how. Foot Ankle Int. 1998 Jan;19(1):52-8. doi: 10.1177/107110079801900111. No abstract available. PMID 9462915